CLINICAL TRIAL: NCT00117962
Title: A Randomized Phase II Study of Radiation Therapy, Pemetrexed and Carboplatin With or Without Cetuximab in Stage III Non-Small Cell Lung Cancer
Brief Title: Pemetrexed Disodium, Carboplatin, and Radiation Therapy With or Without Cetuximab in Treating Patients With Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Eli Lilly and Company (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB 30407; U10CA031946 (NIH); CDR0000434616 (Other: Physician Data Query)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Results first posted 2013-01-15 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Cetuximab; Carboplatin; Pemetrexed; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Std Tx + Pemetrexed (Experimental): Patients receive pemetrexed disodium IV over 10 minutes followed by carboplatin IV over 30 minutes on days 1, 22, 43, and 64. Patients also undergo thoracic radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, 36-40, and 43-47.
  Interventions: Drug: carboplatin; Drug: pemetrexed disodium; Radiation: radiation therapy
- Std Tx + Pemetrexed and Cetuximab (Experimental): Patients receive pemetrexed disodium, carboplatin, and thoracic radiotherapy as in arm I. Patients also receive cetuximab IV over 2 hours on day 1 and then IV over 1 hour on days 8, 15, 22, 29, 36, and 43.
  Interventions: Biological: cetuximab; Drug: carboplatin; Drug: pemetrexed disodium; Radiation: radiation therapy

INTERVENTIONS:
Biological: cetuximab — 400 mg/sq m IV over 120 min: Day 1; Week 1 250 mg/sq m IV over 60 min weekly for 6 more weeks.
  Arms: Std Tx + Pemetrexed and Cetuximab
Drug: carboplatin — AUC = 5 q 21 days for 4 cycles
Drug: pemetrexed disodium — 500 mg/sq m IV q 21 days during chemoradiation and consolidation chemotherapy phases
Radiation: radiation therapy — Thoracic radiotherapy: 70 Gy for 7 weeks beginning on Day 1.

SUMMARY:
RATIONALE: Pemetrexed disodium may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also make tumor cells more sensitive to radiation therapy. Giving pemetrexed disodium, carboplatin, and radiation therapy together with cetuximab may kill more tumor cells.

PURPOSE: This randomized phase II trial is studying how well giving pemetrexed disodium and carboplatin together with radiation therapy with or without cetuximab works in treating patients with stage III non-small cell lung cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the overall survival of patients with unresectable stage III non-small cell lung cancer treated with pemetrexed disodium, carboplatin, and thoracic radiotherapy with or without cetuximab.

Secondary

* Determine the failure-free survival and response rates in patients treated with these regimens.
* Correlate epidermal growth factor receptor, erbB2, and K-ras mutations with survival and tumor response in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study.

* Chemoradiotherapy (courses 1-4): Patients are randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive pemetrexed disodium IV over 10 minutes followed by carboplatin IV over 30 minutes on days 1, 22, 43, and 64. Patients also undergo thoracic radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, 36-40, and 43-47.
  * Arm II: Patients receive pemetrexed disodium, carboplatin, and thoracic radiotherapy as in arm I. Patients also receive cetuximab IV over 2 hours on day 1 and then IV over 1 hour on days 8, 15, 22, 29, 36, and 43.
* Consolidation chemotherapy (courses 5-8): Beginning 3-5 weeks after completion of chemoradiotherapy, all patients receive consolidation chemotherapy comprising pemetrexed disodium alone IV over 10 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 3 years.

PROJECTED ACCRUAL: A total of 100 patients (50 per treatment arm) will be accrued for this study within 10-13 months.

ELIGIBILITY:
1. Histologically or cytologically documented NSCLC, including squamous cell carcinoma, adenocarcinoma including bronchoalveolar cell, and large cell anaplastic carcinoma (including giant and clear cell carcinomas)
2. Eligible Disease Stages: Inoperable IIIA and Selected IIIB - Patients entered must be considered unresectable or inoperable. Patients do not need to have a mediastinoscopy.

   A size of 2 cm or greater by CT is a sufficient criterion for the diagnosis of mediastinal lymph node (N2 or N3) involvement by malignancy. If the largest mediastinal lymph node is less than 2 cm in diameter, a biopsy confirmation of mediastinal nodal involvement is required.
   1. The following patients are eligible:

      * Patients must be M0
      * Patients with any T with N2 or N3 are eligible
      * Patients with T3, N1-N3 disease are eligible if deemed unresectable
      * Patients with T4, any N are eligible provided the T4 status is not determined because of malignant effusion
      * Patients with contralateral mediastinal disease (N3) are eligible if all gross disease can be encompassed in the radiation field in accordance with the homogeneity criteria
      * Patients with a pleural effusion, which is a transudate, cytologically negative and non-bloody, are eligible if the radiation oncologist feels the tumor can be encompassed within a reasonable field of radiotherapy
      * If a pleural effusion can be seen on the chest CT but not on CXR and is too small to tap, the patient will be eligible. Patients who develop a new pleural effusion after thoracotomy or other invasive thoracic procedure will be eligible.
   2. The following patients are NOT eligible:

      * Patients with T3, N0 disease
      * Patients with M1 disease
      * Patients with atelectasis of the entire lung
      * Patients with direct invasion of vertebral body
      * Patients with scalene, supraclavicular, or contralateral hilar node involvement
      * Patients with exudative, bloody, or cytologically malignant effusions
3. Patients must have Measurable Disease: Lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥10 mm with spiral CT scan. Lesions that are not considered measurable include bone lesions, leptomeningeal disease, ascites, pleural/pericardial effusion, abdominal masses that are not confirmed and followed by imaging techniques, cystic lesions and tumor lesions situated in a previously irradiated area.
4. Prior Therapy: ≥ 2 weeks since formal exploratory thoracotomy. No prior chemotherapy for NSCLC, chest radiation therapy or therapy that specifically and directly targets the EGFR pathway
5. ECOG performance status 0-1
6. Positron Emission Tomography (PET) using 18 fluorodeoxyglucose (FDG) must be negative for distant metastasis. PET imaging is mandatory.
7. Weight loss of ≤ 10% in the past 3 months
8. No "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse.
9. Non-pregnant and non-nursing because of significant risk to the fetus/infant
10. Age ≥ 18 years
11. No patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness.
12. No HIV-positive patients receiving combination anti-retroviral therapy because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy
13. No known history of hypersensitivity to carboplatin, pemetrexed or a monoclonal antibody
14. Required Initial Laboratory Values:

    1. Granulocytes ≥ 1,500/mcl
    2. Platelets ≥ 100,000/mcl
    3. Calculated Creatinine Clearance ≥ 45 ml/min
    4. Bilirubin < 1.5 x ULN
    5. AST/ALT < 3 x ULN
    6. Alkaline Phosphatase < 3 x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2005-09; Primary Completion 2009-03 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Govindan, MD, Study Chair — Washington University School of Medicine
Locations (71):
- United States (71):
  - Arroyo Grande Community Hospital, Arroyo Grande, California
  - Eden Medical Center, Castro Valley, California
  - Saint Rose Hospital, Hayward, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Valley Care Medical Center, Pleasanton, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Bendheim Cancer Center at Greenwich Hospital, Greenwich, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Iowa Blood and Cancer Care, Cedar Rapids, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Upper Chesapeake Medical Center, Bel Air, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton MD, Maryland
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Missouri Cancer Associates, Columbia, Missouri
  - Siteman Cancer Center at Barnes-Jewish St. Peters Hospital - Saint Louis, St Louis, Missouri
  - St. Anthony's Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - Saint Francis Cancer Treatment Center at Saint Francis Memorial Health Center, Grand Island, Nebraska
  - Callahan Cancer Center at Great Plains Regional Medical Center, North Platte, Nebraska
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - Mount Sinai Medical Center, New York, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - Southwest Virginia Regional Cancer Center at Wellmonth Health, Norton, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - St. Mary's Regional Cancer Center at St. Mary's Medical Center, Huntington, West Virginia

REFERENCES:
- [Result] Govindan R, Bogart J, Stinchcombe T, Wang X, Hodgson L, Kratzke R, Garst J, Brotherton T, Vokes EE. Randomized phase II study of pemetrexed, carboplatin, and thoracic radiation with or without cetuximab in patients with locally advanced unresectable non-small-cell lung cancer: Cancer and Leukemia Group B trial 30407. J Clin Oncol. 2011 Aug 10;29(23):3120-5. doi: 10.1200/JCO.2010.33.4979. Epub 2011 Jul 11. PMID 21747084

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2005 and January 2008, 109 participants were recruited.
Pre-assignment Details: Six (6) participants cancelled before receiving any protocol related therapy and 2 participants were deemed ineligible; therefore, 101 participants were analyzed.
Period: Overall Study
Arm/Group | Std Tx + Pemetrexed | Std Tx + Pemetrexed and Cetuximab
Started | 48 | 53
Completed | 26 | 28
Not Completed | 22 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Std Tx + Pemetrexed | Std Tx + Pemetrexed and Cetuximab | Total
Number analyzed (Participants) | 48 | 53 | 101
Age, Continuous [Median (Full Range); unit: years] | 65 [41 to 79] | 66 [32 to 81] | 66 [32 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 27 | 34 | 61
Region of Enrollment [Number; unit: participants]
  United States | 48 | 53 | 101
Histology [Number; unit: participants]
  Adenocarcinoma | 22 | 22 | 44
  Squamous | 17 | 18 | 35
  NSCLC, undifferentiated | 8 | 10 | 18
  Large cell | 0 | 2 | 2
  Not reported | 1 | 1 | 2
ECOG Performance Status [Number; unit: participants] — Classifies patients according to their functional impairment. Scores range from 0 (fully active) to 5 (death).
  participants
    0 - Fully Active | 28 | 18 | 46
    1 - Ambulatory, restricted strenuous activity | 20 | 35 | 55
TNM Stage [Number; unit: participants] — American Joint Committee on Cancer, Cancer Staging Manual http://www.cancerstaging.org/products/pasteditions.html
  participants
    IIIA | 29 | 27 | 56
    IIIB | 18 | 24 | 42
    Not reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: 18 Month Survival
Description: Percentage of participants who were alive at 18 months. The 18 month survival, with 95% CI, was estimated using the Kaplan-Meier method.
Time Frame: 18 months (from randomization)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Std Tx + Pemetrexed | Std Tx + Pemetrexed and Cetuximab
Number analyzed (Participants) | 48 | 53
percentage of participants | 58 [46 to 74] | 54 [42 to 70]

2. Secondary Outcome: Failure-free Survival
Description: Failure-free survival (FFS) is the time from randomization to a failure event, defined as disease progression or death from any cause (which ever occurred first). The median FFS with 95% CI was estimated using the Kaplan-Meier method,
Time Frame: Time from randomization to failure (up to 4 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Std Tx + Pemetrexed | Std Tx + Pemetrexed and Cetuximab
Number analyzed (Participants) | 48 | 53
months | 12.6 [7.9 to 17.2] | 12.3 [8.8 to 18.7]

3. Secondary Outcome: Number of Participants With Overall Tumor Response
Description: Response was defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria:
  * Complete Response (CR): disappearance of all target lesions;
  * Partial Response (PR) 30% decrease in sum of longest diameter of target lesions;
  * Progressive Disease (PD): 20% increase in sum of longest diameter of target lesions;
  * Stable Disease (SD): small changes that do not meet above criteria.
  Overall tumor response is the total number of CR and PRs.
Time Frame: Duration of study until progression (up to 4 years)
Measure: Number; unit: participants
Arm/Group | Std Tx + Pemetrexed | Std Tx + Pemetrexed and Cetuximab
Number analyzed (Participants) | 48 | 53
participants | 37 | 38

4. Other Pre Specified Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from patient randomization (arm assignment) to death from any cause. The median OS with 95% CI was estimated using the Kaplan-Meier method.
Time Frame: Time from randomization to death (up to 4 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Std Tx + Pemetrexed | Std Tx + Pemetrexed and Cetuximab
Number analyzed (Participants) | 48 | 53
months | 21.2 [17.5 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment | 25.2 [14.4 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment

ADVERSE EVENTS:
Description: Adverse events were evaluated for 103 participants (50 and 53 on arm A and B, respectively).
Arm/Group | Std Tx + Pemetrexed | Std Tx + Pemetrexed and Cetuximab
Serious Adverse Events (participants affected / at risk) | 21/50 | 25/53
Other Adverse Events (participants affected / at risk) | 48/50 | 50/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Std Tx + Pemetrexed (N=50) | Std Tx + Pemetrexed and Cetuximab (N=53)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 2 (3)
Hemoglobin decreased (Blood and lymphatic system disorders) | 14 (20) | 12 (16)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 3 (3)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (6) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 5 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 8 (13) | 14 (19)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 4 (5) | 0 (0)
Esophageal stenosis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 7 (10) | 8 (10)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 3 (4) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (13) | 6 (7)
Oral pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Proctoscopy abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (9) | 5 (6)
Chest pain (General disorders) | 1 (1) | 3 (3)
Chills (General disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 2 (3)
Fatigue (General disorders) | 17 (27) | 15 (20)
Fever (General disorders) | 5 (5) | 1 (1)
General symptom (General disorders) | 0 (0) | 1 (1)
Localized edema (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (2) | 3 (3)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Phlebitis infective (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Small intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 5 (6)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 5 (5)
Blood bilirubin increased (Investigations) | 3 (3) | 3 (6)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 4 (5) | 2 (2)
INR increased (Investigations) | 2 (2) | 0 (0)
Laboratory test abnormal (Investigations) | 3 (5) | 1 (1)
Leukocyte count decreased (Investigations) | 14 (20) | 18 (27)
Lymphocyte count decreased (Investigations) | 3 (3) | 5 (9)
Neutrophil count decreased (Investigations) | 11 (15) | 14 (21)
Platelet count decreased (Investigations) | 14 (18) | 17 (26)
Serum cholesterol increased (Investigations) | 1 (1) | 0 (0)
Weight loss (Investigations) | 4 (8) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 6 (9) | 10 (11)
Blood glucose increased (Metabolism and nutrition disorders) | 8 (10) | 8 (10)
Dehydration (Metabolism and nutrition disorders) | 9 (11) | 9 (10)
Serum albumin decreased (Metabolism and nutrition disorders) | 7 (8) | 6 (7)
Serum calcium decreased (Metabolism and nutrition disorders) | 5 (5) | 5 (9)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 5 (6) | 3 (7)
Serum magnesium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (5) | 8 (13)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (2) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 5 (5)
Dysgeusia (Nervous system disorders) | 1 (3) | 2 (2)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (4)
Bladder hemorrhage (Renal and urinary disorders) | 0 (0) | 1 (2)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (4)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 1 (2)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 7 (8)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 7 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 10 (15)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (6)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 5 (5) | 6 (6)
Peripheral ischemia (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 2 (2) | 3 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Std Tx + Pemetrexed (N=50) | Std Tx + Pemetrexed and Cetuximab (N=53)
Blood disorder (Blood and lymphatic system disorders) | 2 (4) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 33 (119) | 29 (151)
Lymphatic disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 4 (5)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (3)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Eye disorder (Eye disorders) | 0 (0) | 2 (4)
Vision blurred (Eye disorders) | 3 (4) | 3 (4)
Watering eyes (Eye disorders) | 2 (3) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 20 (50) | 14 (55)
Diarrhea (Gastrointestinal disorders) | 12 (17) | 13 (31)
Dry mouth (Gastrointestinal disorders) | 2 (10) | 1 (4)
Dyspepsia (Gastrointestinal disorders) | 5 (11) | 8 (16)
Dysphagia (Gastrointestinal disorders) | 28 (92) | 34 (113)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1) | 9 (20)
Esophageal mucositis (Gastrointestinal disorders) | 1 (2) | 1 (2)
Esophageal pain (Gastrointestinal disorders) | 4 (9) | 2 (16)
Esophageal stenosis (Gastrointestinal disorders) | 0 (0) | 3 (7)
Esophagitis (Gastrointestinal disorders) | 22 (73) | 21 (44)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (8) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip pain (Gastrointestinal disorders) | 0 (0) | 1 (3)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 6 (9) | 10 (14)
Nausea (Gastrointestinal disorders) | 27 (73) | 24 (67)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 3 (6) | 0 (0)
Salivary gland disorder (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 20 (52) | 22 (44)
Chest pain (General disorders) | 3 (6) | 3 (8)
Chills (General disorders) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 1 (2) | 2 (5)
Fatigue (General disorders) | 43 (248) | 40 (230)
Fever (General disorders) | 6 (6) | 4 (4)
Flu-like symptoms (General disorders) | 0 (0) | 1 (1)
Gait abnormal (General disorders) | 0 (0) | 1 (1)
General symptom (General disorders) | 1 (1) | 0 (0)
Localized edema (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 2 (4) | 3 (4)
Sudden death (General disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (2) | 3 (3)
Bladder infection (Infections and infestations) | 1 (3) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (5)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 7 (8) | 1 (1)
Lip infection (Infections and infestations) | 0 (0) | 1 (6)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0)
Opportunistic infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (5) | 4 (4)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 2 (5) | 2 (2)
Upper respiratory infection (Infections and infestations) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Vaginal infection (Infections and infestations) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (4)
Dermatitis radiation (Injury, poisoning and procedural complications) | 3 (5) | 3 (9)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 4 (11) | 1 (3)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 11 (20) | 14 (30)
Alkaline phosphatase increased (Investigations) | 1 (1) | 7 (17)
Aspartate aminotransferase increased (Investigations) | 8 (15) | 10 (21)
Blood bilirubin increased (Investigations) | 3 (3) | 4 (8)
Creatinine increased (Investigations) | 6 (11) | 6 (11)
INR increased (Investigations) | 1 (1) | 4 (5)
Laboratory test abnormal (Investigations) | 2 (4) | 0 (0)
Leukocyte count decreased (Investigations) | 38 (141) | 45 (132)
Lymphocyte count decreased (Investigations) | 10 (43) | 14 (70)
Neutrophil count decreased (Investigations) | 28 (94) | 37 (97)
Platelet count decreased (Investigations) | 32 (82) | 37 (111)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 10 (30) | 10 (43)
Anorexia (Metabolism and nutrition disorders) | 17 (41) | 23 (130)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Blood glucose increased (Metabolism and nutrition disorders) | 18 (48) | 21 (52)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 9 (10) | 14 (15)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 14 (30) | 20 (55)
Serum calcium decreased (Metabolism and nutrition disorders) | 5 (7) | 9 (13)
Serum calcium increased (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 10 (13) | 11 (17)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (6) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 11 (13) | 11 (19)
Serum potassium increased (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Serum sodium decreased (Metabolism and nutrition disorders) | 10 (16) | 10 (21)
Serum sodium increased (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 5 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 6 (17) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (10) | 1 (1)
Upper extremity dysfunction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 9 (22) | 7 (15)
Dysgeusia (Nervous system disorders) | 7 (15) | 6 (22)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 6 (8) | 6 (8)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 3 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (22) | 9 (28)
Recurrent laryngeal nerve palsy (Nervous system disorders) | 0 (0) | 1 (22)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 4 (6)
Tremor (Nervous system disorders) | 1 (2) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 3 (4) | 3 (14)
Confusion (Psychiatric disorders) | 2 (2) | 2 (3)
Depression (Psychiatric disorders) | 3 (8) | 4 (15)
Insomnia (Psychiatric disorders) | 8 (30) | 9 (28)
Libido decreased (Psychiatric disorders) | 1 (1) | 1 (1)
Hemoglobin urine positive (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 3 (7) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 1 (3) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 3 (10)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (11)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (61) | 22 (71)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 25 (88) | 19 (51)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (4)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (4)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (3)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 10 (18)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheoscopy abnormal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 6 (31)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (47) | 6 (35)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (6)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 5 (9)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3) | 30 (107)
Rash desquamating (Skin and subcutaneous tissue disorders) | 14 (21) | 20 (38)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Hot flashes (Vascular disorders) | 1 (2) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 4 (10) | 4 (4)
Lymphedema (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischemia (Vascular disorders) | 1 (10) | 0 (0)
Phlebitis (Vascular disorders) | 2 (3) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes